CLINICAL TRIAL: NCT00083460
Title: UARK 2001-37, A Phase I Exploratory Study of Combination PS-341 and Thalidomide in Refractory Multiple Myeloma
Brief Title: Study of Combination PS-341 and Thalidomide in Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Brooke Carter, CRA, University_Of_Arkansas
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UARK 2001-37
Record Dates: First submitted 2004-05-24; First posted 2004-05-26 (Estimated); Last update posted 2010-08-02 (Estimated); Status verified 2010-07

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Thalidomide; Velcade; PS-341; Refractory; Bortezomid
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; Thalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: PS-341; Drug: Thalidomide; Drug: Dexamethasone
- 2 (Active Comparator)
  Interventions: Drug: PS-341; Drug: Thalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: PS-341 — Arm 1 a dose of 1.0mg/m2. Arm 2 a dose of 1.3mg/m2
Drug: Thalidomide — In cohort 1, a dose of 50mg for cycles 2-8. Cohort 2, 100mg for cycles 2-8. Cohort 3, 150mg for cycles 2-8. Cohort 4, 200mg for cycles 2-8.
Drug: Dexamethasone — A dose of 20mg for cylces 3-8.

SUMMARY:
The purpose of this study is to assess the toxicity of PS-341 combined with one of four doses of thalidomide in patients with refractory multiple myeloma, and to find the most appropriate doses of PS-341 and thalidomide in the combination.

DETAILED DESCRIPTION:
Patients will be enrolled in groups of 6-10 patients, each receiving a low dose of PS-341 (1.0 mg/m2) and different dose levels of thalidomide (50, 100, 150, and 200 mg). The first six patients in each group will receive PS-341 alone for the first cycle, and thalidomide will be added on day 22. If the combination is found to be safe in these first 6 patients, the remaining patients in each group will be enrolled. Initially, these patients will receive PS-341 alone and thalidomide will be added subsequently, if deemed safe based on the first 6 patients in each thalidomide dose cohort.

ELIGIBILITY:
Inclusion Criteria:

* History of histologically documented multiple myeloma with relapsed or resistant disease, defined as previously treated with/without autologous stem cell transplantation and is either relapsing or is resistant after > 1 line of prior therapy for myeloma
* Patients can not be eligible for MTRC phase III protocols of higher priority
* Performance status of greater than or equal to 2 as per SWOG scale
* Patients must have an absolute neutrophil count > 750/mm3, and a platelet count greater than or equal to 25,000/mm3
* No prior malignancy is allowed except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the patient has been disease free for at least three years. Prior malignancy is acceptable provided there has been no evidence of disease within the three-year interval
* Pregnant or nursing women may not participate. Women of childbearing potential must have a negative pregnancy documented within one week of registration. Women/men of reproductive potential may not participate unless they have agreed to use an effective contraceptive method.
* Male or female adults of at least 18 years of age.
* Signed written informed consent and willingness to meet follow-up schedule and study procedure obligations

Exclusion Criteria:

* Chemotherapy or radiotherapy received within the previous 2 weeks
* Prior Treatment of PS-341
* Significant neurotoxicity, defined as grade greater than or equal to 2 neurotoxicity per NCI Common Toxicity Criteria
* POEMS Syndrome
* Non-secretory multiple myeloma
* Active infection requiring antibiotics
* Clinically significant hepatic dysfunction in the absence of liver metastases as noted by bilirubin or AST >3 times the upper normal limit or clinically significant concurrent hepatitis
* New York Hospital Association (NYHA) Class III or Class IV heart failure
* Myocardial infarction within the last 6 months
* Poorly controlled hypertension, diabetes mellitus, or other serious or psychiatric illness that could potentially interfere with the completion of treatment according to this protocol
* Severe renal dysfunction defined as a creatinine clearance < 20 cc/min.
* Absolute neutrophil count < 750/mm3, and a platelet count < 25,000/mm3
* Pregnant or potential for pregnancy
* Breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2001-12; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Assess the toxicity of PS-341 combined with one of four doses of thalidomide in patients with refractory multiple myeloma | until pt progresses or unexceptible toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Barlogie Barthel, M.D. Ph.D, Principal Investigator — University of Arkanas for Medical Sciences website
Locations (1):
- University of Arkansas for Medical Sciences/MIRT, Little Rock, Arkansas, United States

REFERENCES:
- See also: Myeloma Institute for Research & Therapy website — http://myeloma.uams.edu